CLINICAL TRIAL: NCT04684251
Title: ARTerial EMbolization for haemorrhoIdal Disease Study
Brief Title: ARTerial EMbolization for haemorrhoIdal Disease (ART.EM.I. Study)
Acronym: ARTEMIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding no longer available.
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12397
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Haemorrhoidal Bleeding
Keywords: haemorrhoid; embolisation
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment arm (Experimental): The treatment arm will undergo the intervention with embolisation of their hemorrhoidal arteries. The embolisation will be performed using a standard right femoral puncture and after inserting a 5 Fr introducer sheath. The inferior mesenteric artery will be catheterised using a Simmons catheter (radiofocus-Terumo). The superior rectal arteries will be then catheterized with a rapid transit microcatheter Progreat microcatheter (Radiofocus-Terumo) and embolised with coils. The treatment will include the use of fluoroscopy for which the radiation protection department of Oxford University Hospitals NHS Foundation Trust has been consulted. The technical success of the procedure will be assessed fluoroscopically by achieving stasis of blood flow distally to the site of the embolization. CE marked coils will be used for the embolisation of the arteries feeding the haemorrhoids.
  Interventions: Procedure: Coil embolisation of hemorrhoidal arteries.

INTERVENTIONS:
Procedure: Coil embolisation of hemorrhoidal arteries. — Coil embolisation of hemorrhoidal arteries as previously described.

SUMMARY:
Haemorrhoidal disease is amongst the most common rectal conditions causing significant distress to the affected patients. Current surgical techniques for the treatment of internal haemorrhoids are associated with several drawbacks and sometimes high recurrence rates. The purpose of this study is to assess the safety and efficacy of a new minimally invasive technique that is based on blocking the arteries that feed the haemorrhoids and thus potentially leading to a decrease in their size. A recently published paper with 14 patients showed good results in terms of safety(Vidal et. al.). Despite the promising preliminary evidence, there is still a need for more studies and additional data. Furthermore, at the current time, there are no studies assessing quality of life changes post embolisation for these patients and the investigators hope to evaluate this important aspect of treatment as well.

This study will provide the investigators with results regarding the efficacy and safety of arterial embolisation for advanced haemorrhoid disease. This will be the first study to provide data on short and long term efficacy (in terms of re-bleeding and re-operation rates) as well as to provide evidence on the effect of this novel treatment on quality of life. This study will also be the largest study to date and if successful will pave the way for a large randomised controlled trial comparing the gold standard surgical treatment to the embolisation treatment.

The embolisation of haemorrhoid vessel is not an experimental technique and it has been used in the past in cases of uncontrollable hemorrhoidal- related bleeding with good results and without morbidity. However, this is the first time that the investigators will use this technique as a first line treatment for haemorrhoids and part of this study is to assess the feasibility and safety of this approach.

DETAILED DESCRIPTION:
This is a pilot, prospective, single arm and single centre trial to assess the safety and efficacy of haemorrhoid embolisation. Patients with advanced hemorrhoidal disease (grade II-IV) will be identified through the colorectal clinic with a recruitment target of 24 patients. The duration of patient participation in this study is 24 months. During this time the patient will have to attend 4 appointments (including the treatment session).

All cases in this study will be performed as day case procedures. The patients will be admitted to the interventional radiology day unit in the morning, where a standard pre-assessment will take place. The main intervention will be the embolisation of their hemorrhoidal arteries. The embolisation will be performed using a standard approach with a right femoral puncture and after inserting a 5 Fr introducer sheath. The inferior mesenteric artery will be catheterized using a Simmons catheter (radiofocus-Terumo). The superior rectal arteries will be then catheterized with a rapid transit microcatheter Progreat microcatheter (Radiofocus-Terumo) and then embolised with a number of coils. The arteries will be packed with coils until there is complete blood flow stasis within the target artery bilaterally. The technical success of the procedure will be assessed by achieving stasis of blood flow distally to the site of the embolisation. This will be assessed fluoroscopically. CE marked coils will be used for the embolisation of the arteries feeding the haemorrhoids.

Following the procedure, patients will be discharged to their usual place of residence after 6 hours of observations in the interventional radiology day unit. The patients will be followed up in the colorectal clinic after 3 months, 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

i. Adult male and female patients between the ages of 40-90 years old.

ii. Patients with grade II-IV haemorrhoid disease with re-current or active bleeding AND

iii. Patients with (ii) who do not wish to undergo surgery for their symptoms OR

iv. Patients with (ii) despite previous surgery.

v. Patients who can understand and sign the consent form.

Exclusion Criteria:

i. Patients who are not otherwise fit for surgery.

ii. Patients with significant ano-rectal comorbidities (cancer, fistula, abscesses).

iii. Patients who are unable to sign the inform consent form.

iv. Pregnancy.

v. Patients with history of significant colorectal disease or previous colectomy.

vi. Iodine allergy/ Contrast allergy.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
To assess the clinical success of the procedure | Pre-operative (day of procedure) 3, 12, and 24 months post-operatively
  Resolution of symptoms 1 year after operation is the primary endpoint. This will be assessed with a previously validated patient questionnaire of bowel function (Nyström et. al.). Five questions about haemorrhoidal symptoms will be appended while retaining the structure of the questionnaire. Patients will also submit a health-related quality-of-life questionnaire (SF-12 Form). Questionnaires will be completed before the operation, at 3, 12 and 24 months follow-up.

SECONDARY OUTCOMES:
To assess the technical success of the procedure | Day of procedure (immediately at time of procedure)
  The technical success of the procedure will be assessed by achieving stasis of blood flow distally to the site of the embolization. This will be assessed fluoroscopically.
To assess the safety of the procedure and potential side effects | Immediately post-procedure, 3, 12 and 24 months post-operatively
  Post-operative pain will be recorded by the patient after operation. The pain experienced during most of the day and a peak pain will be recorded straight after the procedure and using a ten point visual analogue scale (VAS) (0, no pain; 10, worst pain imaginable). Side effects and potential complications related to the procedure will be documented in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Raman Uberoi, FRCR, Principal Investigator — John Radcliffe Hospital, Oxford University Hospitals NHS Foundation Trust, Headington, Oxford OX3 9DU
Locations (1):
- Department of Interventional Radiology, John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vidal V, Louis G, Bartoli JM, Sielezneff I. Embolization of the hemorrhoidal arteries (the emborrhoid technique): a new concept and challenge for interventional radiology. Diagn Interv Imaging. 2014 Mar;95(3):307-15. doi: 10.1016/j.diii.2014.01.016. Epub 2014 Feb 28. PMID 24589187
- [Background] Nystrom PO, Qvist N, Raahave D, Lindsey I, Mortensen N; Stapled or Open Pile Procedure (STOPP) trial study group. Randomized clinical trial of symptom control after stapled anopexy or diathermy excision for haemorrhoid prolapse. Br J Surg. 2010 Feb;97(2):167-76. doi: 10.1002/bjs.6804. PMID 20035531